CLINICAL TRIAL: NCT05571176
Title: KetaMoHydBup: Pharmacokinetic Interaction of S-ketamine, Morphine, Hydromorphone and Buprenorphine
Acronym: KetaMoHydBup
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Elina Brinck (Other)
Responsible Party: Sponsor-Investigator, Elina Brinck, MD, PhD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBrinck; 2021-006011-28 (EudraCT Number)
Record Dates: First submitted 2022-09-28; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: The Effect of S-ketamine on Pharmacokinetics of Morphine, Hydromorphone, and Buprenorphine
Keywords: S-ketamine; hepatic UGT2B7 enzyme; pharmacokinetic interaction; morphine; hydromorphone; buprenorphine
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: This is a cross-over study with two phases on 12 healthy volunteers. Study participants will be administered S-ketamine 0.29mg/kg/h intravenously or placebo (NaCl 0.9%) for 4 hours. 30 minutes after the initiation of the study drug infusion, each subject will be given single boluses of morphine 0.01mg/kg, hydromorphone 0.002mg/kg and buprenorphine 0.003mg/kg IV. We will analyze pharmacokinetic parameters (Cmax, tmax, AUC, t1/2) for morphine, hydromorphone, and buprenorphine. The aim of the study is to evaluate whether S-ketamine has a pharmacokinetic interaction with the opioids (morphine, hydromorphone, buprenorphine) known to be metabolized via liver UGT2B7 enzyme.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Study participants, investigators, care providers and personnel collecting samples are blinded. Personnel preparing study drugs will not participate on conducting the study. On the first phase of the study, study participants will be administered one of the study drug infusions (either S-ketamine or placebo). The order of the study drug is random. On the second phase, study participants will be administered the other study drug (S- ketamine or placebo) that she/he did not receive on the first phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine infusion (Experimental): 12 healthy volunteers, S-ketamine infusion 0.29 mg/kg/h for 4 hours
  Interventions: Drug: S-ketamine
- Placebo (NaCl 0.9%) infusion (Placebo Comparator): 12 healthy volunteers, placebo (NaCl 0.9%) infusion for 4 hours
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: S-ketamine — S-ketamine infusion 0.29 mg/kg/h for 4 hours

SUMMARY:
S-ketamine is often administered as a part of multimodal analgesia to reduce postoperative pain and postoperative opioid consumption. Current data indicates that ketamine may be useful for patients with prior use of opioids whereas the benefit for opioid-naive patients is less clear. However, different opioids have variable pharmacokinetic characteristics. Therefore, it is important to evaluate S-ketamine's effect on the pharmacokinetics of opioids.

DETAILED DESCRIPTION:
S-ketamine is often used as a part of multimodal analgesia to reduce postoperative pain and opioid consumption, in part by mitigating opioid tolerance and opioid-induced hyperalgesia. However, there are mixed results concerning the effect of ketamine for this indication. Different opioids have various pharmacokinetic characteristics. Ketamine is known to inhibit the liver UGT2B7-enzyme, that is responsible for e.g., morphine metabolism. Therefore, it is important to investigate whether there is a clinically important pharmacokinetic interaction between S-ketamine and opioids metabolized via liver UGT2B7 enzyme. These opioids include morphpine, hydromorphone and buprenoprhine.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age 18-45 years
* healthy
* Normal values in the following laboratory assessments: Hb, P-ALAT, P-AFOS, P-GT, P-creatinine, P-K, P-Na, chemical sample for urine (U-KemSeul). Pregnancy test (P-hCG-tot) must be negative.
* Urine sample for detection of any illegal drugs must be negative (U-Huum-PS)
* Normal EKG
* Normal blood pressure
* No prior use of illicit drugs

Exclusion Criteria:

* Tendency/predisposition to illicit drug use, illicit drug use in history
* Abnormal EKG
* smoking
* use of oral contraceptives
* pregnancy, lactation
* participating in a less tha 3 months ago
* Blood donation less than 3 months ago
* The subject's peripheral veins are hardly visible (predisposing difficulties in cannulation)
* weight less than 50 kg, body mass index (BMI) less than 18,5 or over 30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of morphine, hydromorphone and buprenorphine after intravenous S-ketamine infusion. | Time points for the measurements after the initiation of S-ketamine infusion: 0 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes and 210 minutes
  We aim to investigate whether there is a clinically significant pharmacokinetic interaction between S-ketamine and morphine, S-ketamine and hydromorphone and S-ketamine and buprenorphine.
Peak plasma concentrations (Cmax) of morphine, hydromorphone and buprenorphine after intravenous S-ketamine infusion | Time points for assessing peak plasma concentrations (Cmax) for morphine, hydromorphone and buprenorphine are the following: 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes, 210 minutes after the initiation of S-ketamine infusion.
  We aim to investigate whether there is a clinically significant pharmacokinetic interaction between S-ketamine, morphine, S-ketamine and hydromorphone and S-ketamine and buprenorphine.
Half-life time (t1/2) of morphine, hydromorphone and buprenorphine concentrations after intravenous S-ketamine infusion. | Time points for assessing half-life time of morphine, hydromorphone and buprenorphine are 0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes and 210 minutes after initiation of S-ketamine infusion.
  We aim to investigate whether there is a clinically significant pharmacokinetic interaction between S-ketamine, morphine, S-ketamine and hydromorphone and S-ketamine and buprenorphine.

SECONDARY OUTCOMES:
The effect of S-ketamine on brain-derived neurotrophic factor (BDNF) release | Time points for assessments: 30 minutes, 120 minutes, 240 minutes, 360 minutes, 480 minutes and at Day1 after the intiation of S-ketamine infusion
  We measure BDNF plasma levels (ng/ml) during and after intravenous S-ketamine infusion .
The effect of S-ketamine on vascular endothelial growth factor (VEGF) release | Time points for assessments: 30 minutes, 120 minutes, 240 minutes, 360 minutes, 480 minutes and at Day1 after the intiation of S-ketamine infusion.
  We measure VEGF levels (ng/l) during and after intravenous S-ketamine infusion.
The effect of S-ketamine infusion on prolactin release. | Time points for assessments: 30 minutes, 120 minutes, 240 minutes, 360 minutes, 480 minutes and at Day1 after the intiation of S-ketamine infusion
  We measure prolactin levels (mU/l) during and after intravenous S-ketamine infusion.
The effect of S-ketamine infusion on cortisol release. | Time points for assessments: 30 minutes, 120 minutes, 240 minutes, 360 minutes, 480 minutes and at Day1 after the intiation of S-ketamine infusion
  We measure cortisol levels (nmol/l) during and after intravenous S-ketamine infusion.
The effect of S-ketamine infusion on thrombocyte aggregation. | At 2 hours after initiation of S-ketamine infusion.
  We evaluate the effect of intravenous S-ketamine infusion on thrombocyte aggregation by using Platelet Function Analyzer (PFA), a method that is based on the property of platelets to adhere upon shear stress conditions and aggregate in consequence of agonist presence in the system. We assess the clotting time. Unit of analysis is seconds (s).

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Lilius, MD, PhD, Principal Investigator — University of Helsinki

IPD SHARING:
Plan to Share IPD: No